CLINICAL TRIAL: NCT02740699
Title: CT COMPARE: CT Coronary Angiography to Measure Plaque Reduction
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Principal Investigator resigned and closed program
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160089; 16-H-0089
Record Dates: First submitted 2016-04-14; First posted 2016-04-15 (Estimated); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2022-03

CONDITIONS: Cardiovascular Disease
Keywords: Cholesterol; Heart Disease; CT Scan; Crestor; Lipitor
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases | interventions — Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Moderate to High Statin Treatment in Participants with Coronary Artery Plaque (Other): Participants with coronary artery plaque will receive moderate to high statin treatment at either 20-40 mg once daily Rosuvastatin or 40-80 mg once daily of Atorvastatin.
  Interventions: Drug: Rosuvastatin; Drug: Atorvastatin; Radiation: Cardiac Computed Tomography (CT); Radiation: Cardiac Magnetic Resonance Image (MRI)

INTERVENTIONS:
Drug: Rosuvastatin — Participants will receive 20-40 mg once daily
  Other Names: Crestor
Drug: Atorvastatin — Participants will receive 40-80 mg once daily.
  Other Names: Lipitor
Radiation: Cardiac Computed Tomography (CT) — Cardiac CT angiography (CCTA) provides a non-invasive method of evaluating both calcified and noncalcified plaque volume. Performed at baseline, 12 months 24 months, and 36 months.
  Other Names: Cardiac CT angiography (CCTA)
Radiation: Cardiac Magnetic Resonance Image (MRI) — Provides a non-invasive method of evaluating both calcified and noncalcified plaque volume. Cardiac MRI may be performed at baseline, and 24 months (optional).
  Other Names: Cardiovascular Magnetic Resonance Imaging (CMR)

SUMMARY:
Background:

Coronary artery disease causes plaque in arteries. This can cause stroke or heart disease. Drugs called statins might shrink plaque. Researchers want to study how CT scanning can determine if an individuals arterial plaque has decreased while taking statins.

Objectives:

To measure the change in coronary artery plaque volume in people treated with high-intensity statin therapy using CT and MRI scans. To study the metabolic activity of plaque in arteries. To determine how well plaque measurements from heart CT scans can be replicated.

Eligibility:

Men ages 40-75 and women ages 40-75 who are good candidates for statin treatment

Design:

Visit 1: participants will be screened with:

* Medical history
* Blood tests
* Heart MRI and CT scan: An IV inserted into an arm or hand vein removes blood and injects contrast, and medicine if needed. Participants lie on a table that slides into a machine that takes pictures of the body. For the CT scan, if their heart rate is too high, they get medicine to lower it. They breathe in a special way, holding their breath for 5 seconds.

Participants will begin high-intensity statin treatment.

Participants will have 7 more visits over 3 years. All visits include blood tests and medication review. Some may also include:

* Statin treatment adjustment
* CT scan
* MRI scan
* Physical exam

Participants may join the PET Substudy. This includes 5 more visits during the study. These include:

* Getting an IV in an arm vein
* Blood tests
* PET scans: They fast 12 hours before.

Participants may join the Reproducibility Substudy if they had a slow heart rate during their first CT scan. This includes 1 additional heart CT scan 4 weeks later.

DETAILED DESCRIPTION:
In high risk patients undergoing invasive angiography, intravascular ultrasound (IVUS) has shown reduction of plaque for patients treated with HMG-CoA reductase inhibitors (statins). However, there is no accepted noninvasive method to determine if treatment for atherosclerosis results in reduction of coronary artery plaque.

Coronary artery CT angiography (CCTA) is noninvasive and can accurately determine the degree of coronary artery stenosis. In addition, the extent of calcified and noncalcified plaque may be directly measured using this technology at low radiation dose using state-of-the-art CT scanners. Several retrospective studies have previously suggested that CCTA may be able to show plaque regression in the coronary arteries due to statin therapy.

The primary aim of this proposal is to determine the change in coronary artery plaque volume in individuals treated with high intensity statin therapy as defined by 2013 ACC/AHA Guideline on the Treatment of Blood Cholesterol to Reduce Atherosclerotic Cardiovascular Risk in Adults.

Men and women who meet the inclusion and exclusion criteria will undergo CCTA examination for the presence or absence of coronary artery plaque. Individuals with evidence of noncalcified coronary plaque by CCTA and who meet criteria for HMG-CoA reductase (statin) therapy will be evaluated for a total of 36 months. The change of coronary artery plaque (progression or no change, or regression) in individuals with noncalcified plaque at baseline will be measured by CCTA at yearly intervals.

ELIGIBILITY:
* INCLUSION CRITERIA:

A. Men greater than or equal to 40 and less than or equal to 75 years of age; women greater than or equal to 40 and less than or equal to 75 years of age

B. Willing to travel to the NIH for follow-up visits.

C. Willing to start or modify statin therapy.

D. Able to understand and sign informed consent.

E. Eligible for primary prevention statin therapy

1. Eligible for at least moderate intensity statin according to 2013 ACC/AHA GRCR (i.e., greater than or equal to 5% 10 year cardiovascular risk, https://my.americanheart.org/professional/StatementsGuidelines/Prevention-Guidelines_UCM_457698_SubHomePage.jsp) OR
2. low (<5%) 10 year cardiovascular risk per 2013 ACC/ AHA and with coronary artery calcium score greater than or equal to 300 Agatston units or greater than or equal to 75 percentile for age, sex, and ethnicity determined per MESA study

(http://www.mesa-nhlbi.org/calcium/input.aspx).

EXCLUSION CRITERIA:

A. Allergy or prior clinically relevant adverse reaction to Rosuvastatin (does not include minor muscle pain).

B. High intensity statin treatment for more than 90 days prior to enrollment

C. LDL greater than or equal to 190 mg/ml

D. Physician-diagnosed heart attack

E. Physician-diagnosed stroke or TIA

F. Physician-diagnosed heart failure

G. Having undergone procedures related to cardiovascular disease (CABG, angioplasty, valve replacement, pacemaker or defibrillator implantation, any surgery on the heart or arteries)

H. Active treatment for cancer

I. Prior hypersensitivity reaction to iodinated contrast injection

J. Known hyperthyroidism.

K. Acute renal failure, renal transplant, dialysis and renal failure clinically diagnosed.

L. History of liver transplant or severe liver disease or unexplained elevation of baseline ALT>3x upper limit of normal

M. Pregnancy and nursing

N. Mental, neurologic or social condition preventing understanding of the rationale, procedures, risks and potential benefits associated with the trial.

O. Any other conditions that precludes safety for MRI and/or CT imaging per the researcher's evaluation.

P. Individuals with hemoglobinopathies or severe asthma.

Q. Severe renal excretory dysfunction, estimated glomerular filtration (eGFR) rate < 30 mL/min/1.73m2 body surface area according to the Modification of Diet in Renal Disease criteria Glomerular filtration rate will be estimated using the MDRD 2005 revised study formula: eGFR (mL/min/1.73m2) = 175 x (standardized serum creatinine)-1.154 x (age)-0.203 x 0.742 (if the subject is female) or x 1.212 (if the subject is black)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nehal N Mehta, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] D'Ascenzo F, Agostoni P, Abbate A, Castagno D, Lipinski MJ, Vetrovec GW, Frati G, Presutti DG, Quadri G, Moretti C, Gaita F, Zoccai GB. Atherosclerotic coronary plaque regression and the risk of adverse cardiovascular events: a meta-regression of randomized clinical trials. Atherosclerosis. 2013 Jan;226(1):178-85. doi: 10.1016/j.atherosclerosis.2012.10.065. Epub 2012 Nov 6. PMID 23206978
- [Background] Ridker PM, Pradhan A, MacFadyen JG, Libby P, Glynn RJ. Cardiovascular benefits and diabetes risks of statin therapy in primary prevention: an analysis from the JUPITER trial. Lancet. 2012 Aug 11;380(9841):565-71. doi: 10.1016/S0140-6736(12)61190-8. PMID 22883507
- [Background] Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2889-934. doi: 10.1016/j.jacc.2013.11.002. Epub 2013 Nov 12. No abstract available. PMID 24239923
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-H-0089.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moderate to High Statin Treatment in Participants With Coronary Artery Plaque
Started | 79
Completed | 55
Not Completed | 24
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 14
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | Moderate to High Statin Treatment in Participants With Coronary Artery Plaque
Number analyzed (Participants) | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 49
Age, Continuous [Mean (Full Range); unit: years] | 65.4 [48.7 to 75.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 78
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 72
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 79

OUTCOME MEASURES:

1. Primary Outcome: Mean Change of Non-calcified Plaque Volume in Participants Treated With High Intensity Statin Therapy Assessed by Coronary Computed Tomography Angiography
Description: Mean change of non-calcified plaque volume assessed by Coronary computed tomography angiography in participants treated with high intensity statin therapy (as defined by the 2013 ACC/AHA Guidelines to Reduce Cardiovascular Risk (GRCR).
  Using anatomical landmarks, a target plaque volume will be defined at baseline and follow up examinations. Software will be used to trace lumen and outer vessel boundaries to determine non-calcified plaque volume.
  The 2013 ACC/AHA Guidelines to GRCR focuses on the assessment of cardiovascular risk, lifestyle modifications to reduce cardiovascular risk and management of elevated blood cholesterol and body weight in adults. High-intensity statin therapy is defined by: rosuvastatin 20-40 mg or atorvastatin 40-80 mg. The maximum statin dose will be administered that is tolerated by the patient and that maintains LDL-C > or = 25 mg/dl. High-intensity statin therapy is defined as lowering LDL-C on average by approximately > or = 50%.
Time Frame: Baseline and 24 months
Population: Intention to treat analysis for those participants with observed plaque volumes by Coronary artery CT angiography at baseline and 24 months will be included in the primary analysis.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Moderate to High Statin Treatment in Participants With Coronary Artery Plaque
Number analyzed (Participants) | 55
mm^3 | 23.3 (76.6)
Statistical Analysis 1: Comparison: Moderate to High Statin Treatment in Participants With Coronary Artery Plaque; Test type: Superiority; p = 0.0256, Wilcoxon Signed Rank Tests

2. Secondary Outcome: Mean Change of Non-calcified Plaque Volume in Participants Treated With High Intensity Statin Therapy Assessed by Coronary Computed Tomography Angiography
Description: as for outcome 1
Time Frame: Baseline and 36 months
Population: Intention to treat for those participants with observed plaque volumes by Coronary artery CT angiography at baseline and 36 months will be included in the secondary analysis.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Moderate to High Statin Treatment in Participants With Coronary Artery Plaque
Number analyzed (Participants) | 52
mm^3 | 8.86 (75.3)
Statistical Analysis 1: Comparison: Moderate to High Statin Treatment in Participants With Coronary Artery Plaque; Test type: Superiority; p = 0.0254, Wilcoxon Signed Rank Tests

3. Secondary Outcome: Linear Mixed-effects Regression Coefficient of Age Effect on Plaque Volume
Description: Linear mixed-effects regression coefficient of age effect on plaque volume measured by Coronary artery CT angiography. Plaque volumes (mm3) were quantified from coronary CTA exams using a validated automated method developed by Cleerly. Regression coefficient is the mean change of plaque volume given one year increase of age. In the mixed-effects model the outcomes are plaque volumes measured at Baseline, 24 months and 36 months as described in 2011 "Applied Longitudinal Analysis" Wiley Series in Probability and Statistics by Fitzmaurice, Laird, and Ware.
Time Frame: Baseline, 24 months and 36 months
Population: Intention to treat for those participants with observed plaque volumes by Coronary artery CT angiography at baseline, 24 months and 36 months will be included in the secondary analysis.
Measure: Mean (Standard Deviation); unit: mm^3/year
Arm/Group | Moderate to High Statin Treatment in Participants With Coronary Artery Plaque
Number analyzed (Participants) | 52
mm^3/year | 1.48 (2.65)
Statistical Analysis 1: Comparison: Moderate to High Statin Treatment in Participants With Coronary Artery Plaque; Test type: Superiority; p = 0.58, Regression, Linear

4. Secondary Outcome: Linear Mixed-Effects Regression Coefficient of Sex Effect on Plaque Volume (Beta Coefficient)
Description: Linear Mixed-effects Regression Coefficient of sex (female = 0 and male = 1) effect on plaque volume measured by Coronary artery CT angiography (beta coefficient). Plaque volumes (mm3) were quantified from coronary CTA exams using a validated automated method developed by Cleerly. Regression coefficient is the mean change of plaque volume comparing male verses female (female =0 and male = 1). In the mixed-effects model the outcomes are plaque volumes measured at Baseline, 24 months and 36 months as described in 2011 "Applied Longitudinal Analysis" Wiley Series in Probability and Statistics by Fitzmaurice, Laird, and Ware.
Time Frame: Baseline, 24 months and 36 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beta coefficient [mm^3]
Arm/Group | Moderate to High Statin Treatment in Participants With Coronary Artery Plaque
Number analyzed (Participants) | 52
beta coefficient [mm^3] | 100.58 (51.99)
Statistical Analysis 1: Comparison: Moderate to High Statin Treatment in Participants With Coronary Artery Plaque; Test type: Superiority; p = 0.06, Regression, Linear

5. Secondary Outcome: Linear Mixed-effects Regression Coefficient of Race Effect on Plaque Volume (Beta Coefficient)
Description: Linear Mixed-effects Regression Coefficient of Effects race (white = 1 and non-white = 0) effect on plaque volume measured by Coronary artery CT angiography. Plaque volumes (mm3) were quantified from coronary CTA exams using a validated automated method developed by Cleerly. Regression coefficient is the mean change of plaque volume comparing race (white = 1 and non-white = 0). In the mixed-effects model the outcomes are plaque volumes measured at Baseline, 24 months and 36 months as described in 2011 "Applied Longitudinal Analysis" Wiley Series in Probability and Statistics by Fitzmaurice, Laird, and Ware.
Time Frame: Baseline, 24 months and 36 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Beta coefficient [mm^3]
Arm/Group | Moderate to High Statin Treatment in Participants With Coronary Artery Plaque
Number analyzed (Participants) | 52
Beta coefficient [mm^3] | 35.66 (859.39)
Statistical Analysis 1: Comparison: Moderate to High Statin Treatment in Participants With Coronary Artery Plaque; Test type: Superiority; p = 0.69, Regression, Linear

6. Secondary Outcome: Linear Mixed-effects Regression Coefficient of Body Mass Index Effect on Plaque Volume
Description: Linear Mixed-effects Regression Coefficient of Body Mass Index Effect on Plaque Volume measured by Coronary artery CT angiography. Plaque volumes (mm3) were quantified from coronary CTA exams using a validated automated method developed by Cleerly. Regression coefficient is the mean change of plaque volume given one kg/m^2 increase of BMI. In the mixed-effects model the outcomes are plaque volumes measured at Baseline, 24 months and 36 months as described in 2011 "Applied Longitudinal Analysis" Wiley Series in Probability and Statistics by Fitzmaurice, Laird, and Ware.
Time Frame: Baseline, 24 months and 36 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm^3/[kg/m^2]
Arm/Group | Moderate to High Statin Treatment in Participants With Coronary Artery Plaque
Number analyzed (Participants) | 52
mm^3/[kg/m^2] | 7.65 (2.68)
Statistical Analysis 1: Comparison: Moderate to High Statin Treatment in Participants With Coronary Artery Plaque; Test type: Superiority; p = 0.006, Regression, Linear

ADVERSE EVENTS:
Time Frame: Up to 36 months
Arm/Group | Moderate to High Statin Treatment in Participants With Coronary Artery Plaque
All-Cause Mortality (participants affected / at risk) | 0/79
Serious Adverse Events (participants affected / at risk) | 8/79
Other Adverse Events (participants affected / at risk) | 56/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate to High Statin Treatment in Participants With Coronary Artery Plaque (N=79)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Coronary stent placement (Cardiac disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Knee replacement (Surgical and medical procedures) | 1 (1)
Subaraschnoid hemorrhage (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate to High Statin Treatment in Participants With Coronary Artery Plaque (N=79)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Chronic lymphocytic leukemia (Blood and lymphatic system disorders) | 1 (1)
Varicosities (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Systolic murmur (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 7 (9)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Abdominal infection (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Edema limbs (General disorders) | 4 (4)
Fatigue (General disorders) | 2 (3)
Flu like symptoms (General disorders) | 1 (1)
Shoulder pain (General disorders) | 1 (1)
Malaise (General disorders) | 2 (2)
H.pylori (Infections and infestations) | 1 (1)
Lip infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 10 (16)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 11 (14)
Blood bilirubin increased (Investigations) | 3 (5)
CPK increased (Investigations) | 3 (3)
Cholesterol high (Investigations) | 3 (3)
Creatinine increased (Investigations) | 8 (12)
Hyperkalemia (Investigations) | 5 (7)
Hypertriglyceridemia (Investigations) | 8 (14)
Hyponatremia (Investigations) | 5 (7)
Hemoglobin A1C increased (Investigations) | 1 (1)
LDL decreased (Investigations) | 6 (7)
Lymphocyte count decreased (Investigations) | 8 (8)
Lymphocyte count increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 5 (5)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 2 (3)
White blood cell decreased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 17 (17)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (7)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 8 (14)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 5 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Gout attack (Musculoskeletal and connective tissue disorders) | 1 (1)
Prostatitis attack (Musculoskeletal and connective tissue disorders) | 1 (1)
Right Iliotibial band syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Degenerative disc disease (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nodule in Right Lower Lobe (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Concussion (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Foaming urine (Renal and urinary disorders) | 1 (1)
Stage III Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Erythematous plaque and patches (Skin and subcutaneous tissue disorders) | 1 (1)
Hip replacement (Surgical and medical procedures) | 1 (1)
Hot flashes (Vascular disorders) | 1 (3)
Hypertension (Vascular disorders) | 14 (18)
Hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Protocol was terminated early due to departure of Principal Investigator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/99/NCT02740699/Prot_SAP_000.pdf